CLINICAL TRIAL: NCT04679857
Title: Substitution of the Posterior Cruciate Ligament in Total Knee Arthroplasty With Ultracongruent Insert or Posterior Stabilzed Design
Brief Title: Substitution of the PCL in TKA With UC or PS Design
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKA UC PS
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Patient Reported Outcome; Knee Osteoarthritis; Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC (Experimental): Total Knee Arthroplasty with an ultracongruent insert
  Interventions: Other: TKA
- PS (Active Comparator): Total Knee Arthroplasty with posterior stabilized design
  Interventions: Other: TKA

INTERVENTIONS:
Other: TKA — Total Knee Arthroplasty

SUMMARY:
RCT comparing UC and PS TKA

DETAILED DESCRIPTION:
RCT comparing TKA with either ultraconguent insert or posterior stabilized design for substitution of the posterior cruciate ligament

ELIGIBILITY:
Inclusion Criteria:

* scheduled for TKA

Exclusion Criteria:

* higher constraint needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
ROM | 10 years
  Range of motion
Patient reported outcome | 10 years
  Oxford Knee Score min 0 points (worst), max 48 points (best)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Lützner, Principal Investigator — University Hospital Carl Gustav Carus, TU Dresden
Locations (1):
- University Center of Orthopaedics and Traumatology, University Medicine Carl Gustav Carus Dresden, TU Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No